CLINICAL TRIAL: NCT02146859
Title: Predictor of Residual Neuromuscular Blockade in Recovery Room After General Anesthesia
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chaowanan Khamtuikrua, Instructor, Mahidol University
Other Study IDs: Si123
Record Dates: First submitted 2014-05-16; First posted 2014-05-26 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Residual Neuromuscular Blockade
Keywords: residual neuromuscular blockade
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- general anesthesia: Patient having general anesthesia

SUMMARY:
Background When general anesthesia was performed, neuromuscular blocking agents (NMBAs) are frequently used for facilitate tracheal intubation and keep patient still and relax during surgery. Unfortunately, residual neuromuscular blockade are important complication.

There are many factors that affect neuromuscular blockade and may prolong effect of NMBAs which we already know about that such as body temperature, drugs, some kind of diseases. However there are no recent studies that mention about other factors. The purpose of this study is to find out other factors that affect NMBAs effect to improve patient safety.

Methods The study is a prospective, non-randomized, blinded, observational study.

222 patients will be included in this study and will be performed general anesthesia. Anesthetic technique and agent which are used depend on regular staff. Information of patient will be collected are age, sex, weight, height, ASA classification, anesthetic technique, anesthetic and surgical time, amount of inhalation agent, amount of NMBAs, amount of opioids and reversal agents.

After anesthesia finish, patient will be brought to recovery room and Train Of Four watch® will be placed and record Train Of Four ratio by this research staff. Train Of Four ratio < 0.9 will be defined as there is residual neuromuscular blockade in this patient.

All patients will be divided into 2 groups: residual blockade group(patient who have train of four <0.9 after surgery) and no residual blockade group(patient who have train of four >0.9). All factor of each group will be compared between. Statistical will be analyzed to find significant factor which affect neuromuscular blockade.

DETAILED DESCRIPTION:
study about residual neuromuscular blockade

ELIGIBILITY:
Inclusion Criteria:

* - age ≥ 18 years
* American society of anesthesiologist class I-III
* patient who are schedule for intraabdominal surgery, orthopedic surgery and gynecologic surgery under general anesthesia and use neuromuscular blocking agents (NMBAs)

Exclusion Criteria:

* - patients who have myasthenia gravis, myotonia, muscular dystrophy, upper motor neuron lesion
* patients who have drug which influence neuromuscular action such as oral muscle relaxant, anticonvulsants, magnesium sulfate
* Body temperature >37.8 or < 36 degree Celsius before operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient who are schedule for general anesthesia and use neuromuscular blocking agents (NMBAs)
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
residual neuromuscular blockade after surgery | 1 hour
  residual neuromuscular blockade after surgery measure by train of four of nervestimulator

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Siriraj hospital, Bangkok, Thailand